CLINICAL TRIAL: NCT06919354
Title: POLARIS: A Phase 1, Single Dose, Open-label Study of GNTI-122 in Adults With Recently Diagnosed Type 1 Diabetes (T1D)
Brief Title: A Study of GNTI-122 in Adults Recently Diagnosed With T1D
Acronym: POLARIS
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: GentiBio, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GNTI-122-T1D-1001
Record Dates: First submitted 2025-03-25; First posted 2025-04-09 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Type 1 Diabetes (T1D); Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- GNTI-122 (Experimental)
  Interventions: Biological: GNTI-122

INTERVENTIONS:
Biological: GNTI-122 — GNTI-122 is an investigational cell therapy manufactured from a participant's own blood cells and is intended to help correct an imbalance of certain types of cells found in participants with Type 1 Diabetes.

SUMMARY:
This is a 78-week single arm, multi-center, Phase 1 study to evaluate the safety, tolerability, cellular kinetics, and biomarker changes in C-peptide over time of GNTI-122, an investigational cell therapy manufactured from a participant's own blood cells in adult participants with recently diagnosed T1D. After assessment of eligibility, participants who qualify for the study will be enrolled sequentially in 1 of 3 cohorts. Cohort 1 participants (n=3) receive a low dose of GNTI-122 . Cohort 2 participants (n=3) receive a high dose of GNTI-122. Cohort 3 participants (n=10) receive a high dose of GNTI-122 in combination with rapamycin. Participants are followed for 78 weeks after the administration of GNTI-122 during which safety and efficacy assessments are made, including vital signs, ECG, physical exam, clinical labs, and monitoring of adverse events and concomitant medications. Disease markers (e.g., MMTT-stimulated C-peptide, HbA1c) and pharmacodynamic activity (e.g., lymphocyte subsets and phenotypes, effector T cell responses to islet antigens ex vivo, T1D autoantibodies) will be monitored serially throughout the study. The study will include sentinel dosing and a Safety Review Committee to ensure participant safety. Visit https://www.polarisstudy.com to learn more!

DETAILED DESCRIPTION:
This is a 78-week single arm, multi center, Phase 1 study to evaluate the safety, tolerability, cellular kinetics, and biomarker changes in C-peptide over time of GNTI-122 in adult participants with recently (within 120 days of Screening) diagnosed T1D. GNTI-122 is an investigational cell therapy manufactured from a participant's own blood cells and is intended to help correct an imbalance of certain types of cells found in patients with Type 1 Diabetes (T1D).

After assessment of eligibility, participants who qualify for the study will be enrolled sequentially in 1 of 3 cohorts. Cohorts 1 and 2 are safety run-in cohorts (n=3 participants per cohort) in which each participant receives a single dose of GNTI 122 alone; Cohort 1 receives a low dose 1 of GNTI-122 and Cohort 2 receives a high dose of GNTI-122. Cohort 3 includes 10 participants that will receive a single high dose of GNTI-122 in combination with rapamycin (with a target trough concentration [Ctrough] of 3 to 6 ng/mL), which may extend the survival of GNTI-122. Participants will remain at the clinical site for observation for at least 4 hours after administration of GNTI-122.

Safety and tolerability assessments over the 78-week study include: vital signs, 12-lead electrocardiograms, physical examinations, clinical laboratory evaluations, monitoring of adverse events and concomitant medications. Risks to participants will be minimized by the incorporation of sentinel dosing (i.e., at least 28 days of safety assessments between first and second participant and at least 14 days between the second and third participant in Cohorts 1 and 2, and at least 28 days between the first and second participant and the second and third participant in Cohort 3) and the evaluation of safety and tolerability by a Safety Review Committee with at least 14 days of safety assessments (i.e., laboratory values and adverse event reporting) after 3 participants are dosed in Cohort 1 and Cohort 2. Disease markers (e.g., MMTT-stimulated C-peptide, HbA1c) and pharmacodynamic activity (e.g., lymphocyte subsets and phenotypes, effector T cell responses to islet antigens ex vivo, T1D autoantibodies) will be monitored serially throughout the study.

In Cohort 3, rapamycin concentrations will be measured periodically to ensure levels are in the target range of Ctrough level between 3 and 6 ng/mL.

Per Health Authority guidelines (Food and Drug Administration) for gene therapy products or advanced medicinal products, all participants treated with GNTI-122 who complete or discontinue from this study must be monitored for specific toxicities for a total of 15 years (semi-annually or annually), irrespective of their response to GNTI-122. This will be addressed in a separate protocol of a long-term follow-up study of these participants.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female participants aged ≥18 to ≤45 years with recently diagnosed (within 120 days of Screening) T1D according to American Diabetes Association criteria.
2. Participant has residual β-cell function during Screening, defined as random C-peptide ≥ 0.2 nmol/L.
3. Positive for at least one T1D-associated autoantibody.
4. Able and willing to provide written, informed consent as approved by the IRB.
5. Is confirmed positive for the HLA-DRB1*04:01 allele.
6. Has adequate vascular access to undergo leukapheresis with no known contraindications.

8. Female participants of childbearing potential must have a negative serum pregnancy test at Screening, must be not lactating, and must agree to protocol-specified contraception.

9. Male participants of childbearing potential must agree to protocol specified contraception.

10. Other than T1D, participant is in good general health.

Exclusion Criteria:

1. Type 2 diabetes.
2. Experienced DKA within 4 weeks prior to or during Screening.
3. Unwilling or unable to comply with study procedures or schedule.
4. Chronic or uncontrolled medical condition.
5. Has another active or autoimmune or inflammatory disease with the exception of well-controlled Hashimoto's thyroiditis, celiac disease, or vitiligo.
6. Participation in another clinical study or active follow-up in a prior study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2025-09-03 (Actual); Primary Completion 2028-02 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability of GNTI-122 with and without rapamycin in adult participants with recently diagnosed T1D | Week 78
  Cumulative AEs/SAEs and clinically significant abnormalities in physical exams, vital signs, clinical laboratory measures, and other clinical assessments

SECONDARY OUTCOMES:
Cellular kinetics of GNTI-122 with and without rapamycin in adult participants with recently diagnosed T1D | Week 78
  Measurement of maximum concentration of circulating engineered regulatory T cells as measured by droplet digital polymerase chain reaction
Cellular kinetics of GNTI-122 with and without rapamycin in adult participants with recently diagnosed T1D | Week 78
  Measurement of area under the concentration-time curve [AUC] of circulating engineered regulatory T cells
Cellular kinetics of GNTI-122 with and without rapamycin in adult participants with recently diagnosed T1D | Week 78
  Measurement of half-life of circulating engineered regulatory T cells

CONTACTS AND LOCATIONS:
Overall Officials: Mark Bach, MD, Study Director — GentiBio, Inc
Locations (10):
- United States (10):
  - City of Hope Medical Center, Duarte, California
  - University of California - San Diego, San Diego, California
  - University of California - San Francisco, San Francisco, California
  - University of Florida - Gainesville, Gainesville, Florida
  - University of Miami, Diabetes Research Institute, Miami, Florida
  - Joslin Diabetes Center, Boston, Massachusetts
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Columbia University, New York, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Duke University, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: Yes
Sponsor will share study results via a publication or conference presentation.

REFERENCES:
- See also: For more information, see our POLARIS study website — https://www.polarisstudy.com/